CLINICAL TRIAL: NCT07407335
Title: Effect of Teach-Back Breastfeeding Education on Breastfeeding Success, Breastfeeding Self-Efficacy, and Mother-Infant Bonding in Primiparous Postpartum Women: A Randomized Controlled Trial
Brief Title: Teach-Back Breastfeeding Education After Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nilgun Avci (Other)
Responsible Party: Sponsor-Investigator, Nilgun Avci, phD, Biruni University
Organization: Biruni University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Teach-Back Breastfeeding
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breastfeeding; Postpartum Period
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach-Back Breastfeeding Education (Experimental): Participants received standard postpartum breastfeeding education plus an additional teach-back session delivered one time at postpartum 3-4 hours. The session lasted approximately 30 minutes in total, including education and participant feedback. Content included key elements of effective breastfeeding (latch, audible swallowing, nipple type, breast/nipple comfort, and positioning/hold) and signs of successful breastfeeding.
  Interventions: Behavioral: Teach-Back Breastfeeding Education
- Control: Standard Breastfeeding Education (No Intervention): Participants received standard postpartum breastfeeding education routinely provided by the hospital (lactation nurse-led), without a teach-back component.

INTERVENTIONS:
Behavioral: Teach-Back Breastfeeding Education — Participants received standard postpartum breastfeeding education plus an additional teach-back session delivered one time at postpartum 3-4 hours. The session lasted approximately 30 minutes in total, including education and participant feedback. Content included key elements of effective breastfeeding (latch, audible swallowing, nipple type, breast/nipple comfort, and positioning/hold) and signs of successful breastfeeding.
  Arms: Teach-Back Breastfeeding Education

SUMMARY:
This study evaluated whether breastfeeding education delivered using the teach-back method improves breastfeeding outcomes and mother-infant bonding among primiparous postpartum women. Early postpartum breastfeeding education is routinely provided in many hospitals; however, women may have difficulty remembering or applying the information after birth. Teach-back is a communication method where the patient is asked to explain the information back in their own words, allowing the educator to check understanding and clarify misconceptions.

In this randomized controlled trial, postpartum women who gave birth in a private hospital were assigned either to a teach-back breastfeeding education group or to a control group receiving standard breastfeeding education. Breastfeeding success, breastfeeding self-efficacy, and mother-infant bonding were assessed using validated measurement tools at postpartum 6 hours and again at postpartum 24 hours.

The findings of this study aim to support evidence-based postpartum breastfeeding education practices and improve early breastfeeding outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women who gave birth at the study hospital during the study period
* Primiparous postpartum women
* Live birth
* Volunteered to participate and provided informed consent

Exclusion Criteria:

* Multiparous women
* Neonatal or perinatal loss
* Mothers who refused breastfeeding
* Inability to communicate in Turkish
* Hearing impairment or mental health conditions limiting participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Success | At postpartum 6 hours and postpartum 24 hours
  Breastfeeding success assessed using the LATCH Breastfeeding Assessment Tool.

SECONDARY OUTCOMES:
Breastfeeding Self-Efficacy | At postpartum 6 hours and postpartum 24 hours
  Breastfeeding self-efficacy assessed using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF).
Mother-Infant Bonding | At postpartum 6 hours and postpartum 24 hours
  Mother-infant bonding assessed using the Mother-to-Infant Bonding Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- State Obstetrics and Gynecology Hospital, Istanbul, Bayrampaşa, Istanbul, Turkey (Türkiye)